CLINICAL TRIAL: NCT03833297
Title: Monitoring the HePAtological TOXicity of Drugs
Brief Title: Monitoring the HePAtological TOXicity of Drugs (HePATOX)
Acronym: HePATOX
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-19-02
Record Dates: First submitted 2019-02-04; First posted 2019-02-07 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Liver Diseases; Liver Dysfunction; Liver Failure; Hepatotoxicity
Keywords: hepatological disease; hepatotoxicity; chemotherapies; drugs
MeSH Terms: conditions — Liver Diseases; Liver Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Hepatological toxicity induced by drugs and chemotherapies: Case reported in the World Health Organization (WHO) of hepatological toxicities of patient treated by a drug, with a chronology compatible with the drug toxicity
  Interventions: Drug: Drugs inducing hepatological toxicity

INTERVENTIONS:
Drug: Drugs inducing hepatological toxicity — Drugs susceptible to induce hepatological toxicities

SUMMARY:
Several drugs and chemotherapies seem to have an impact on the hepatological system. This study investigates reports of hepatological toxicities, including the International classification of disease ICD-10 for treatments in the World Health Organization (WHO) global Individual Case Safety Report (ICSR) database (VigiBase).

DETAILED DESCRIPTION:
Several drugs and chemotherapies seem to have an impact on the hepatological system and are responsible of a wide range of hepatological diseases and side effects. Those are poorly described, due to the modification of the pharmacopeia, and the recent recognition of several of these adverse events. This study investigates the main characteristics of patients affected by rare hepatological side effects imputed to drugs. A causality assessment according to the WHO-UMC (World Health Organization - Uppsala Monitoring Center) is systematically applied.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the WHO's pharmacovigilance database till 04/02/2019

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a drug that could be reported in the WHO's pharmacovigilance database
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Hepatological toxicities of drugs Identification and report of cases of hepatological toxicities associated with drugs. | Case reported in the World Health Organization (WHO) database of individual safety case reports to 04/02/2019

SECONDARY OUTCOMES:
Causality assessment of reported hepatological toxicities events according to the WHO system | Case reported in the World Health Organization (WHO) database of individual safety case reports to 04/02/2019
Description of the type of hepatoilogical toxicity depending on the category of drug | Case reported in the World Health Organization (WHO) database of individual safety case reports to 04/02/2019
Description of the other immune related adverse events concomitant to the hepatological toxicity induced by drugs | Case reported in the World Health Organization (WHO) database of individual safety case reports to 04/02/2019
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | Case reported in the World Health Organization (WHO) database of individual safety case reports to 04/02/2019
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) database of individual safety case reports to 04/02/2019
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) database of individual safety case reports to 04/02/2019
Description of the population of patients having hepatological toxicity adverse event | Case reported in the World Health Organization (WHO) database of individual safety case reports to 04/02/2019

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided